CLINICAL TRIAL: NCT05984602
Title: A Phase IB Study to Determine the Safety and Tolerability of Canakinumab and Tislelizumab in Combination With Nab-Paclitaxel and Gemcitabine in the Neo-adjuvant Treatment of Patients With Pancreatic Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-01205
Record Dates: First submitted 2023-08-02; First posted 2023-08-09 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer, GI cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Gastrointestinal Neoplasms | interventions — canakinumab; tislelizumab; 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Quadruplet regimen prior to resection for pancreatic cancer (Experimental): Treatment of Canakinumab and Tislelizumab in Combination with Nab-Paclitaxel and Gemcitabine up to 4 cycles (4 months)
  Interventions: Drug: Canakinumab; Drug: Tislelizumab; Drug: Nab-Paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: Canakinumab — 250 mg subcutaneous injection in prefilled syringes on day 1 of every 28-day cycle
  Other Names: ACZ885
Drug: Tislelizumab — 300 mg in a liquid vial (concentrate for intravenous (i.v.) solution) on day 1 of every 28-day cycle
Drug: Nab-Paclitaxel — 125 mg/m2 intravenous infusion on days 1, 8, 15 of every 28-day cycle
Drug: Gemcitabine — 1000 mg/m2 intravenous infusion on days 1, 8, 15 of every 28-day cycle

SUMMARY:
The goal of this Single Arm Phase Ib clinical trial is to test standard of care chemotherapy and anti PD1 and IL1b to evaluate the safety and preliminary toxicity of this quadruplet regimen prior to resection in patients with pancreatic cancer. The main objectives it aims to answer are to:

* Determine the recommended Phase II dose regimen of canakinumab and tislelizumab in combination with gemcitabine and nab-paclitaxel in patients with localized pancreatic ductal adenocarcinoma.
* Estimate the proportion of patients who proceed to surgical resection.
* Determine the safety and tolerability of canakimumab in combination with tislelizumab, nab-paclitaxel and gemcitabine
* Assess the preliminary clinical anti-tumor activity of canakimumab in combination with tislelizumab, nab-paclitaxel and gemcitabine
* Assess whether therapy has any impact on surgical options

Participants will have labs drawn, CT scans, and a treatment administered consisting of:

* Gemcitabine
* Nab-paclitaxel
* Canakinumab
* Tislelizumab

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years at the time of informed consent
* Histologically or cytologically confirmed pancreatic ductal adenocarcinoma (PDAC) as determined by a local laboratory (adenosquamous is also allowed).
* Tumor confined to the pancreas and deemed resectable or borderline resectable per NCCN guidelines for these criteria.
* Patients must have not received previous anti-cancer therapy for the treatment of pancreatic ductal adenocarcinoma.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Adequate organ function (laboratory results must be obtained within the 21-day screening window) including hematologic, renal and hepatic function.

  * Absolute neutrophil count > 1500/mm3
  * Platelets > 100,000/mm3
  * Calculated creatinine clearance > 60 mL/min (Cockcroft Gault)
  * Albumin > 3.0 g/dL
  * Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT) serum glutamic pyruvic transaminase (SGPT) < 3.0 x ULN
  * Total bilirubin ≤ 1.5 X ULN
* Able to adhere to study visit schedule and other protocol requirements
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study therapy
* Female subjects of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity for the course of the study through 9 months after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year

Exclusion Criteria:

* - Diagnosis of pancreatic neuroendocrine carcinoma or pancreatic acinar cell carcinoma.
* Determined by the medical or surgical team to be a poor candidate for future surgical resection
* Has locally advanced or metastatic disease as determined by imaging

  o This includes those with a baseline CA 19-9 level > 1000 as these subjects have a high rate of metastatic disease
* Previous immunotherapy (e.g. anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways) for pancreatic cancer.
* Known microsatellite instability-high (MSI-H) or mismatch repair-deficient pancreatic cancer
* Any prior treatment with canakinumab or drugs of a similar mechanism of action (IL-1 inhibitor).
* Administration of a live vaccine within 30 days of the first dose of therapy on study
* History of known hypersensitivity to any of the drugs used in this study or any of their excipients, or patient has contraindication to any of the study drugs as outlined in the local prescribing information (e.g. United States Prescribing Information [USPI])
* Active autoimmune disease that has required systemic treatment in the past 2 years prior to enrollment i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs. Control of the disorder with replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is permitted.
* Patient has concurrent malignancy other than the disease under investigation, with exception of malignancy that was treated curatively and has not recurred within 2 years prior to the date of screening. Fully resected basal or squamous cell skin cancers, and any carcinoma in situ are eligible.
* Subjects with a history of pneumonitis or interstitial lung disease requiring therapy
* Patient with suspected or proven immunocompromised state or infections, including:

  * Evidence of active or latent tuberculosis (TB) as determined by locally approved screening methods. If the results of the screening per local treatment guidelines or clinical practice require treatment, then the patient is not eligible.
  * Known history of testing positive for Human Immunodeficiency Virus (HIV) infections.
  * Any other medical condition (such as active infection, treated or untreated), which in the opinion of the investigator places the patient at an unacceptable risk for participation in immunomodulatory therapy.

Note: Patients with localized condition unlikely to lead to a systemic infection e.g. chronic nail fungal infection are eligible.

* Pre-existing peripheral neuropathy > Grade 1 (CTCAE V 5.0)
* Allogeneic bone marrow or solid organ transplant
* Uncontrolled or severe cardiac disease. e (history of unstable angina, myocardial infarction, coronary stenting, or bypass surgery within the prior 6 months), symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia [including atrial flutter/fibrillation], requirement for inotropic support or use of devices for cardiac conditions [pacemakers/defibrillators]), uncontrolled hypertension defined by a systolic blood pressure =>160 mg and/or diastolic blood pressure =>100 mg Hg.
* Any significant medical condition, laboratory abnormality or psychiatric condition that would constitute unacceptable safety risks to the patients, contraindicate patient participation in the clinical study, limit the patient's ability to comply with study requirements, or compromise patient's compliance with the protocol and all requirements of the study as stated in the Informed Consent Form.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-07-14 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of dose limiting toxicities (DLTs) | 56 days
  A dose-limiting toxicity (DLT) is defined as an adverse event (AE) or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first 8 weeks of study treatment. NCI CTCAE v5.0 will be used for all grading.
Number of patients who proceeded to surgical resection | End of treatment (up to 6 months)
  The study team will collaborate with the surgical team to review whether there are any delays or change in outcome in surgery that is attributed to study drug.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 6 months post treatment
  ORR is defined as the proportion of subjects with best overall response (BOR) of complete response (CR) or partial response (PR), according to RECIST 1.1.
R0 resection rate (R0) | At surgery post treatment (up until 6 months)
  R0 is defined by a surgery that completely removes the visible tumor and that is deemed to be margin negative on final pathology report. If tumor is not completely removed this is will be deemed to have failed to achieve an R0 resection.
Progression Free Survival (PFS) | Up to 6 months after patients last treatment
  PFS is defined as the time from the date of first dose to the date of the first documented disease progression based on local investigator assessment as per RECIST 1.1 (assessed by investigator) or death due to any cause.
Overall Survival (OS) | Up to 6 months after patients last treatment
  OS is defined as the time from date of first dose of study treatment to date of death due to any cause. If a subject is not known to have died, then OS will be censored at the latest date the subject was known to be alive (on or before the cut-off date).
Number of delays outcome of surgery that is attributed to study drug | At surgery post treatment (up until 6 months)
  The surgical team will review whether there are any delays in outcome in surgery that is attributed to study drug.
Number of changes in outcome of surgery that is attributed to study drug | At surgery post treatment (up until 6 months)
  The surgical team will review whether there are any change in outcome in surgery that is attributed to study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Oberstein, MD, Principal Investigator — Perlmutter New York University Cancer Center
Locations (3):
- United States (3):
  - Ambulatory Care Center, New York, New York
  - Clinical Cancer Center, New York, New York
  - NYU Langone Ambulatory Care Center East 38th Street, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: to Paul.Oberstein@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request .Requests should be directed to Paul.Oberstein@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.